CLINICAL TRIAL: NCT00768924
Title: CopiOs(TM) Bone Void Filler in the Post-Harvest Iliac Crest
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 2006-012
Record Dates: First submitted 2008-10-03; First posted 2008-10-08 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2009-02

CONDITIONS: Spinal Fusions
Keywords: Bone Void Filler; Post-Harvest Iliac Crest; Ability of CopiOs to fill the post-harvest iliac crest bone void created by a surgeon during spinal fusion.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Spinal fusion patients

SUMMARY:
The CopiOs Bone Void Filler (BVF) is a synthetic bone graft material consisting of calcium phosphate dehydrate within lyophilized type I bovine collagen that has been formed into pads of various sizes for surgical implantation. Pre-clinical animal studies suggest that the bone healing strength of CopiOs to be equivalent to autograft.

DETAILED DESCRIPTION:
Purpose of the study is to evaluate the in-vivo use of CopiOs bone void filler in a single site trial, providing pre and post-operative evaluations of subjects undergoing spinal fusion with autogenous bone graft, in whom the CopiOs has been used as a bone void filler in the post-harvest iliac crest.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years and older
* Patient must be an appropriate candidate for iliac crest bone harvesting during a spinal fusion.
* Patient must be skeletally mature.
* Patient has signed an IRB approved Informed Consent and HIPAA compliant waiver.

Exclusion Criteria:

* Patient is suffering from any co-morbidities that would excessively increase the risk of surgery, including but not limited to pulmonary or cardiac conditions.
* Patient is pregnant.
* Patient has a severe degenerative bone disease.
* Patient has systemic conditions which would affect bone or wound healing.
* Patient is unwilling or unable to follow postoperative instructions or cooperate in a follow-up program.
* Patient is suffering from mental illness, alcohol abuse or drug abuse.
* Patient has known allergies to bovine collagen.
* Patient has a history of multiple allergies.
* Patient has infection at the surgical site.
* Significantly impaired vascularity proximal to surgical site.
* Sites are in direct contact with articular space.
* Sites where stresses on void will exceed the load strength of fixation hardware.
* Patient has hypercalcemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CopiOs will be used to fill the bony deficit as a result of iliac crest autograft harvest during spinal fusion surgery.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Data obtained by this study will provide valuable insight on the ability of CopiOs to fill the post-harvest iliac crest bone void created by a surgeon during spinal fusion. | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- South Texas Spine Clinic, San Antonio, Texas, United States